CLINICAL TRIAL: NCT01765166
Title: Continuing the Research and Development of Parent Treatment for Child Social Adjustment
Brief Title: Parent Treatment for Child Social Adjustment
Acronym: SSGRIN-PG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019396; 2R44MH065718-04 (NIH)
Record Dates: First submitted 2012-12-17; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Interpersonal Relations
Keywords: Social Skill Training; Social Interaction; Peer relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control(ChO) (Experimental): Children receive traditional SSGRIN child treatment with no parent involvement
  Interventions: Behavioral: SSGRIN-Parent Guide
- Parent attention control(PAC) (Experimental): Children will participate in traditional SSGRIN treatment, and parents will participate in a weekly support group to meet with other parents regarding their child's peer relations and behavior. The support group will meet for a parallel amount of time (1 hour/week for 10 weeks) and be facilitated by two parents with no SSGRIN or Parent Guide experience. The PAC condition will reflect the social support functions of a parenting group, but no therapeutic skills training or other instructional materials will be provided.
  Interventions: Behavioral: SSGRIN-Parent Guide
- Parent Guide-Home Study(PG-HS) (Experimental): Children will receive traditional SSGRIN treatment, and parents will receive the Parent Guide to SSGRIN training by participating in the online Parent Guide Home Study (PG-HS) course. The PG-HS course will include all instructional content and materials for the in-person Parent Guide course, but parent will receive the training online.
  Interventions: Behavioral: SSGRIN-Parent Guide
- Parent Guide(PG) (Experimental): Children will receive traditional SSGRIN treatment and parents will receive parallel traditional in-person SSGRIN-Parent Guide treatment.
  Interventions: Behavioral: SSGRIN-Parent Guide

INTERVENTIONS:
Behavioral: SSGRIN-Parent Guide — All children will receive traditional SSGRIN(Social Skills Group Intervention), but parents will vary in the level of parent treatment. Families will be randomly assigned to one of four treatment conditions(approximately 25% each): (a) Traditional SSGRIN child treatment with no parent involvement (ChO), (b) SSGRIN child treatment plus parent attention control (PAC), (c) SSGRIN child treatment plus Parent Guide-Home-study treatment (PG-HS), or (d) SSGRIN child treatment plus traditional Parent Guide treatment (PG).

SUMMARY:
This Competing Renewal project continues the research and development of a parent-focused intervention, Parent Guide to SSGRIN, which parallels an established child-focused intervention [Social Skills GRoup INtervention (S.S. GRIN); for children ages 8-12 years], in order to teach and reinforce the same social skills and concepts within the home environment. A primary goal is to address questions of relative impact, longer-term treatment benefits, and differential treatment effects of the Parent Guide training on children's social skill development across settings and populations.

DETAILED DESCRIPTION:
This Competing Renewal project continues the research and development of a parent-focused intervention, Parent Guide to SSGRIN, which parallels an established child-focused intervention [Social Skills GRoup INtervention (S.S. GRIN); for children ages 8-12 years], in order to teach and reinforce the same social skills and concepts within the home environment. A primary goal of this Competing Renewal is to conduct a rigorous, large-scale, longitudinal research project that is adequately powered to address questions of relative impact, longer-term treatment benefits, and differential treatment effects of the Parent Guide training on children's social skill development across settings and populations. Though schools often struggle with how to increase parent involvement in school-based programs, school officials report that it is infeasible for them to conduct the full series of in-person parent training groups as the Parent Guide's current curriculum demands; therefore, a second goal of this Competing Renewal is to test a Home-study version of the Parent Guide to bridge training into the home environment. The Home-study version of the Parent Guide will be included as a separate treatment condition within the effectiveness trial. This clinical trial will provide S.S.GRIN treatment for 240 children ages 8-12 and vary the level of parent intervention to determine the effectiveness of the two variations of Parent Guide to S.S.GRIN. Parents will be randomly assigned to one of four conditions: (1) Parent Guide treatment; (2) Parent Guide-Home Study treatment; (3) parent attention control; or (4) no treatment. Pre-treatment, post-treatment, 6-month post-treatment, and 12 month post-treatment data will be collected assessing children's social skill development from children, parents, and teachers. Based on past clinical experience, the probability of adverse psychological and behavioral effects from behavioral intervention is very low; however, to ensure participants' safety, a data and safety monitoring plan will be in place.

ELIGIBILITY:
Inclusion Criteria:children ages 8-12 experiencing peer difficulties who are English speaking. To confirm eligibility regarding peer difficulties, 3-C staff will conduct a brief (5 minute) phone-survey with parents for two sub-scales of the Social Skills Rating System: Parent Form (SSRS; Gresham & Elliott, 1990). To be eligible for participation, a child must have a standard score either (a) less than one standard deviation (std) on the Social Skills Scale (<84%ile) or (b) greater than one std on the Problem Behavior Scale (>84%ile).

-

Exclusion Criteria:SSGRIN group therapy is not recommended for extremely aggressive children (DeRosier, 2005), so any child scoring higher than two std on the Externalizing Problem Behavior Scale (>97%ile) will be excluded from participation and referral sources to other appropriate community resources will be given to parents.

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Children's social skills | pre-treatment, post-treatment, 6 months post-treatment, 12 months post-treatment
  Child Acquired Learning Questionnaire

SECONDARY OUTCOMES:
Parental, child, and dyadic behavioral observations | pre-treatment, post-treatment, 6 months post-treatment, 12 months post-treatment
  Parent-child social problem solving assessment

CONTACTS AND LOCATIONS:
Overall Officials: Melissa E DeRosier, Ph.D., Principal Investigator — 3-C Institute for Social Development; Amanda W Harrell, Ph.D., Principal Investigator — 3-C Institute for Social Development; Allan K Chrisman, M.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - 3-C Institute for Social Development, Cary, North Carolina
  - Duke Child and Family Study Center, Durham, North Carolina

REFERENCES:
- [Background] DeRosier ME. Building relationships and combating bullying: effectiveness of a school-based social skills group intervention. J Clin Child Adolesc Psychol. 2004 Mar;33(1):196-201. doi: 10.1207/S15374424JCCP3301_18. PMID 15028553
- [Background] DeRosier ME, Marcus SR. Building friendships and combating bullying: effectiveness of S.S.GRIN at one-year follow-up. J Clin Child Adolesc Psychol. 2005 Mar;34(1):140-50. doi: 10.1207/s15374424jccp3401_13. PMID 15677288
- [Background] DeRosier, M.E. & Gilliom, M. (2007). Effectiveness of a parent training program for improving children's social behavior. Journal of Child and Family Studies, 16, 660-670.
- [Background] DeRosier, M.E. (1995). Summary of 3-C Program Results with 3rd through 5th graders in the WCPSS.
- [Background] DeRosier, M.E. (2002). Group interventions and exercises for enhancing children's communication,cooperation, and confidence. Sarasota, FL: Professional Resources Press.
- [Background] DeRosier, M.E. (2006). Social Skills Group Intervention - Parent Guide(S.S.GRIN-PG). Cary, NC: SELmedia,Inc.
- See also: 3-C ISD website — http://www.3cisd.com/